CLINICAL TRIAL: NCT02981550
Title: Infection Detection by Breath Analysis
Status: Withdrawn | Type: Observational
Why Stopped: 2 NaNose devices provided inconsistent results in lab calibration testing
Sponsor: BreathTec Biomedical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro18602
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Infection, Community-Acquired; Communicable Disease; Respiratory Infection
Keywords: Infection
MeSH Terms: conditions — Community-Acquired Infections; Communicable Diseases; Respiratory Tract Infections; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled Breath
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this feasibility study is to test a device which analyzes breath and may allow doctors and health professionals to immediately determine if an ill patient has a specific type of bacterial infection. This will allow a health professional to provide immediate targeted antibiotics to properly start treatment without delay.

DETAILED DESCRIPTION:
Community acquired, or hospital acquired [nosocomial] infections [pathogens] are a common cause for morbidity and mortality. Initiation of antibiotic treatment is by best guess or using a broad spectrum antibiotic. The improper administration of antibiotics is known to lead to the developing specter of antibiotic resistant organisms.

Certain community acquired bacterial infection such as Streptococcus upper respiratory tract infections carry increased risk of morbidity secondary to risk of developing abscess, glomerulonephritis, and/or rheumatic fever. Commonly, most upper respiratory tract infections are caused by viruses. However due to the unknown pathogen causing an upper respiratory tract infection, with the risks of potential chronic severe complications from Streptococcus, initial treatment starts with either an antibiotic, or a typical 3day wait for bacterial culture result. Quite often, the wait-and-see approach in the community is not undertaken because of the difficulty in returning for a follow-up appointment.

The risk of a developing antibiotic resistant bacteria is well-known and is one of the greatest health threats worldwide leading to longer hospitalizations, higher medical costs and death, according to the World Health Organization. Thus a point of care device which would enable physicians or other medical practitioners to promptly discriminate between Streptococcal or other antibiotic sensitive pathogens versus non antibiotic sensitive viral causes of specific upper respiratory tract infectious pathogens is needed.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to participate in this study
* Availability of signed informed consent
* Healthy, not on any medication
* Able to provide a breath sample
* Having a condition (eg. suspected strep throat, MRSA, C difficile) which would require a swab/sample for culture

Exclusion Criteria:

* Under the age of 6years
* Eating food or drink (excluding water) within 2 hours of breath test time
* Pregnant or Breastfeeding
* Chronic Obstructive Pulmonary Disease (COPD)
* Inability to comply with study procedure/unable to follow directions
* Currently taking antibiotics or other medication (excluding analgesics)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of Infection detected by exhaled breath analysis confirmed by laboratory culture | Within 3 to 7 days of obtaining culture and exhaled breath sample

CONTACTS AND LOCATIONS:
Overall Officials: Raj Attariwala, MD PhD, Study Director — BreathTec Biomedical Inc.; Yazdan Mirzanejad, MD, Principal Investigator — Fraser Health/University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Junger M, Vautz W, Kuhns M, Hofmann L, Ulbricht S, Baumbach JI, Quintel M, Perl T. Ion mobility spectrometry for microbial volatile organic compounds: a new identification tool for human pathogenic bacteria. Appl Microbiol Biotechnol. 2012 Mar;93(6):2603-14. doi: 10.1007/s00253-012-3924-4. Epub 2012 Feb 12. PMID 22327321
- [Background] Thorn RM, Greenman J. Microbial volatile compounds in health and disease conditions. J Breath Res. 2012 Jun;6(2):024001. doi: 10.1088/1752-7155/6/2/024001. Epub 2012 May 4. PMID 22556190
- [Background] Bos LD, Sterk PJ, Schultz MJ. Volatile metabolites of pathogens: a systematic review. PLoS Pathog. 2013 May;9(5):e1003311. doi: 10.1371/journal.ppat.1003311. Epub 2013 May 9. PMID 23675295